CLINICAL TRIAL: NCT01839721
Title: Impact of Probiotics BIFILACT® on Diarrhea in Patients Treated With Pelvic Radiation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Mimi Demers, registered dietitian, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5.7.06.09
Record Dates: First submitted 2013-04-16; First posted 2013-04-25 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Cancer; Diarrhea; Abdominal Pain; Quality of Life
Keywords: Probiotics; radiation-induced enteritis; radiation-induced diarrhea; radiation, diarrhea, enteritis; diet; nutrition
MeSH Terms: conditions — Neoplasms; Diarrhea; Abdominal Pain; Enteritis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bifilact® probiotics standard dose (Active Comparator): concentration of 1.3 billion of Lactobacillus acidophilus LAC-361 and Bifidobacterium longum BB-536. one pill twice a day. Each capsule contained maltodextrin and magnesium stearate as excipient
  Interventions: Drug: Bifilact®
- Bifilact® probiotics high dose (Active Comparator): containing 10 billion Lactobacillus acidophilus LAC-361 and Bifidobacterium longum BB-536. One pill three times a day. Each capsule contained maltodextrin and magnesium stearate as excipient
  Interventions: Drug: Bifilact®
- placebo (Placebo Comparator): Each capsule contained maltodextrin and magnesium stearate as excipient. One pill twice a day
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Bifilact® — placebo, standard dose 1.3 billion twice a day, high dose 10 billion three time a day
  Other Names: probiotics
  Arms: Bifilact® probiotics high dose; Bifilact® probiotics standard dose
Other: placebo
  Arms: placebo

SUMMARY:
In this double-blinded randomized clinical trial study, investigators assessed probiotic used to prevent or delay radiation induced grade moderate to severe diarrhea with patient treated for pelvic cancer.

DETAILED DESCRIPTION:
This study was prospective, unicentric, controlled with comparison to a placebo, randomised and double-blinded. Patients were stratified into three groups: prostatic cancers, gynecologic cancers without chemotherapy and gynecologic or rectal cancers with chemotherapy.

Patients were block-randomized by the research nurse and received a standard dose of Bifilact® probiotics or placebo according to the random list generated by blocks of 2, 4, or 6 patients according to random permutations. A preliminary internal pilot study was performed when the half of the expected sample size were recruited. The goal of this analysis was to test assumptions that lead to chosen sample sizes (N0) and thus, validate the feasibility of the study. Following preliminary results, the sample size re-calculated at the interim analysis is similar to that originally intended. It would be advisable to continue the recruitment as planned. No adjustment to the critical level of the test would be required in analyzes carried out at the end of study. However, another random block using higher probiotics dosage to the randomization was added with preservation of double bind. New random list were generated for each strata with a 3:1:1 ratio (higher dose, standard dose, placebo) to compensate for the starting of the latest higher dose group. All the bottles had a similar aspect, they were all identified by the commercial brand Bifilact. Also the group, either A, B or C, was circled on that bottle, depending on if that bottle belong to the placebo group, standard dose group, or high dose group. Only the nurse knew the coding system, it was also her who would assign the patient to a group, according to the randomization list. She would also hand out the bottle to the patient every week. The two registered dietician, caregivers, were totally excluded of this processes (preliminary study and randomisation) to preserve the double blind.

ELIGIBILITY:
Inclusion Criteria:

* They had a pelvic cancer: gynecologic, rectal, or prostatic,they were to receive radiotherapy treatments for a minimum of 40 Gy at the pelvic level , with or without chemotherapy and they had Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1

Exclusion Criteria:

* they had previous radiotherapy treatments in the pelvic or abdominal region, medical history of gastro-intestinal inflammation, malabsorption syndrome or inflammatory bowel disease or coeliac disease, ileostomy, daily use of anti-diarrheal medication before radiotherapy, pregnancy or breastfeeding, neutropenia or probiotics intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2006-12; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
testing the efficacy of probiotics Bifilact®, in comparison to a placebo to assess its ability to prevent or delay the incidence of moderate or severe symptoms of diarrhea during the period of treatment by radiotherapy | day 1-60
  Patients were asked to note in a daily logbook whether they experienced digestive problems such as daily bowel movements. Severity of the diarrhea was evaluated according to toxicity criteria of the WHO: grade 1 = increase of 2-3 stools per day compared to pre-treatment, grade 2 = increase of 4-6 bowel stools per day or nocturnal stools, grade 3 = increase of 7-9 stools per day or incontinence, grade 4 = increase of 10 or more stools, need for IV hydration. The Registered Dietitian assessed symptoms in logbook with the patient once a week.The duration of daily logbook was 4-9 weeks depending of the total dose of external radiotherapy

SECONDARY OUTCOMES:
Secondary objectives were to assess whether intake of Bifilact® lowered the interruption of radiotherapy treatments or doses of both radiotherapy or chemotherapy | week 1-9
  Registered Dietitian assessed respect of the preview protocol treatment each week (radiotherapy and chemotherapy) if not respected: diarrhea is it involved. For patients that received chemotherapy, a weekly blood profile was obtained and study pills were discontinued if neutrophil count became ≤1.5 X 10(9)/L.
Secondary objective were to assess whether intake of Bifilact® decreased or delayed the consumption of anti-diarrheal medication | day 1-60
  Patients were asked to note, each day during the treatment,in a daily logbook intake of anti-diarrheal medication, laxatives, and antibiotics. The Registered Dietitian assessed symptoms noted with the patient each week.The duration of daily logbook was 4-9 weeks depending of the total dose of external radiotherapy
Secondary objectives were to assess whether intake of Bifilact® reduced abdominal pain | day 1-60
  Abdominal pain was evaluated according to the NCI scale version 3.0: Grade 1 = mild pain, not interfering with function, grade 2 = moderate pain: pain or analgesics interfering with function, but not interfering with activity of daily living, grade 3 =: severe pain: pain or analgesics severely interfering with activity of daily living. The Registered Dietitian assessed information with the patient each week
Secondary objectives were to assess whether the overall well-being of patients was improved during treatment. | week 0, 4-9, 6-11
  Quality of life (EORTC-QLQ-C30) assessment was filled three times during the study: once at the outset, once at the end, and then again two weeks after the last radiotherapy treatment.
Secondary objectives were to assess whether intake of Bifilact® decreased need for hospitalization | week 1-9
  Registered Dietitian assessed each week if the patient had need hospitalization and if the diarrhea has involved

CONTACTS AND LOCATIONS:
Overall Officials: Dagnault Anne, PhD, Study Director — CHU de Quebec; Josee Desjardins, B.Sc, RD, Principal Investigator — Chu de Quebec; Mimi Demers, B.Sc. RD, Principal Investigator — CHU de Québec
Locations (1):
- CHU de Québec, radio-oncology departement, Québec, Quebec, Canada

REFERENCES:
- [Derived] Demers M, Dagnault A, Desjardins J. A randomized double-blind controlled trial: impact of probiotics on diarrhea in patients treated with pelvic radiation. Clin Nutr. 2014 Oct;33(5):761-7. doi: 10.1016/j.clnu.2013.10.015. Epub 2013 Oct 24. PMID 24200199